CLINICAL TRIAL: NCT07014397
Title: Effect of Oral Valaciclovir on Inter- Appointment Endodontic Pain in Single-Rooted Necrotic Teeth With Symptomatic Apical Periodontitis: A Randomized Clinical Trial
Brief Title: Effect of Valaciclovir on Inter-Appointment Pain in Endodontic Treatment of Necrotic Teeth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IR.TUMS.DENTISTRY.REC.1403.045
Record Dates: First submitted 2025-06-02; First posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2024-06

CONDITIONS: Symptomatic Apical Periodontitis
Keywords: symptomatic apical periodontitis (SAP); herpes viruse; pain; valacyclovir
MeSH Terms: conditions — Pain | interventions — Valacyclovir

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- placebo group (Placebo Comparator)
  Interventions: Drug: Placebo
- valacyclovir group (Experimental)
  Interventions: Drug: Valacyclovir

INTERVENTIONS:
Drug: Valacyclovir — valacyclovir group received 2 g (two 1 g tablets) one hour prior to treatment, followed by 2 g 12 hours later, and 1 g at both 24 and 36 hours post-treatment
  Arms: valacyclovir group
Drug: Placebo — The control group received a placebo identical in appearance and administration schedule
  Arms: placebo group

SUMMARY:
Aim: To investigate the effect of oral valacyclovir on inter-appointment endodontic pain in single-rooted necrotic teeth diagnosed with symptomatic apical periodontitis (SAP).

Materials and Methods: This study was a randomized, triple-blind, placebo-controlled clinical trial conducted on 38 teeth. Participants were assigned to intervention or control groups using stratified randomization based on gender and baseline pain severity. Both groups received similar root canal treatment; the only difference was the administration of valacyclovir in the intervention group and placebo in the control group. Patients' pain levels were monitored and recorded at 6, 24, and 48 hours post-treatment using a Visual Analog Scale (VAS), along with their consumption of analgesic (ibuprofen).

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 60 years of age
* Require primary root canal treatment (RCT) in single-rooted maxillary or mandibular teeth (anterior or posterior)
* Diagnosed with symptomatic apical periodontitis (SAP) with confirmed pulp necrosis

Exclusion Criteria:

* Teeth with unrestorable crowns
* Presence of endodontic-periodontal or pure endodontic lesions
* Complex root canal anatomies as defined by the AAE Endodontic Case Difficulty Assessment Form
* Internal or external root resorption
* Calcified canals
* Root canal configuration other than Vertucci's Type I
* Pain originating from more than one tooth
* Marginal periodontitis
* Parafunctional habits
* Systemic diseases classified as ASA class II or higher
* Diagnosed migraine or other headache disorders mimicking orofacial pain
* Intellectual or cognitive impairments
* Pregnancy or breastfeeding
* Use of medications affecting pain perception
* Current use of antibiotics or antiviral agents
* Known allergies to study medications

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-03-22 (Actual); Study Completion 2025-03-26 (Actual)

PRIMARY OUTCOMES:
Pain intensity measured by Visual Analog Scale (VAS) | 6, 24, and 48 hours post-treatment
  The Visual Analog Scale (VAS) is a commonly used tool for assessing pain intensity in patients. In this method, the patient is asked to indicate the perceived level of pain on a 10-centimeter horizontal line, where 0 represents "no pain" and 10 denotes "the worst pain imaginable." Based on the scores provided by patients, pain intensity is categorized into three levels: scores from 0 to 3 indicate mild pain, 4 to 7 indicate moderate pain, and 8 to 10 indicate severe pain.

SECONDARY OUTCOMES:
Proportion of participants requiring ibuprofen as rescue analgesic | Within 48 hours post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Adnaninia, DDS, Principal Investigator — Tehran University of Medical Sciences
Locations (1):
- Tehran University of Medical Sciences, School of Dentistry, Tehran, Iran

IPD SHARING:
Plan to Share IPD: Undecided